CLINICAL TRIAL: NCT04785677
Title: Multisite Randomized Controlled Trial of Comprehensive Trauma Informed Reentry Services for Moderate to High Risk Youth Releasing From State Prisons
Brief Title: Researching Resiliency in Stressful Experiences (RISE) Program for Men Leaving Incarceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen Tripodi, Professor;, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001064; 2019-MU-CX-0065 (Other Grant/Funding Number: National Institute of Justice)
Record Dates: First submitted 2021-02-05; First posted 2021-03-08 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Stress Disorders, Traumatic; Stress Disorders, Traumatic, Acute; Depressive Symptoms; Anxiety; Substance Use; Aggression; Coping Skills; Impulsive Behavior; Housing Problems; Recidivism; Stress; Occupational Stress; Psychological Distress
Keywords: employment stability; Housing Stability; Reentry; Trauma; psychological wel-being
MeSH Terms: conditions — Stress Disorders, Traumatic; Stress Disorders, Traumatic, Acute; Depression; Anxiety Disorders; Substance-Related Disorders; Aggression; Impulsive Behavior; Recidivism; Occupational Stress; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Trauma-Based Reentry Program (Experimental): Participants will complete up to19 session comprehensive trauma-based reentry program.
  Interventions: Behavioral: Resiliency in Stressful Experiences (RISE) Program
- Treatment as usual (TAU) (No Intervention): Participants will be receive all reentry services normally eligible to receive by the state or the community to which they are released.

INTERVENTIONS:
Behavioral: Resiliency in Stressful Experiences (RISE) Program — The Resiliency in Stressful Experiences (RISE) Program is a multi-phased comprehensive trauma based reentry program designed based on the transitional nature of reentry. Participants will receive up to 4 sessions prior to release and up tp 15 session post release from prison. The RISE program is a trauma intervention paired with reentry services, including housing support and employment assistance.
  Other Names: Comprehensive Trauma-Based Reentry Program
  Arms: Comprehensive Trauma-Based Reentry Program

SUMMARY:
The investigators are conducting a randomized controlled trial to assess the impact of Resiliency in Stressful Experiences (RISE) - a comprehensive trauma-based program for young men releasing from a southeastern state's prisons. The investigators are assessing whether treating trauma and providing other transitional supports - such as employment assistance - as young men return home will help to improve their community stability and enhance their psychological well-being, in turn, resulting in less likelihood that a person will become incarcerated in the future.

DETAILED DESCRIPTION:
The five-year study is a two-armed, randomized controlled trial evaluating the effectiveness of a comprehensive trauma-based reentry program for young men assessed as moderate to high risk for recidivism as they are released to the community. Four Hundred young males who were released from one of ten Florida prisons into our target counties were randomly assigned to receive a comprehensive trauma-based reentry program or treatment as usual. The effectiveness of the reentry program was evaluated on mechanisms of change (trauma symptoms, coping, impulsivity, and aggression), community stability (housing, employment), and recidivism.

Research questions are: Does a comprehensive trauma-based research program improve key mechanisms of change for moderate to high-risk young males? Does a comprehensive trauma-based reentry program improve community stability for moderate to high-risk young males? Does a comprehensive trauma-based reentry program decrease rates of recidivism for moderate to high-risk young males? Research questions 1 and 2 were analyzed using ANCOVA, and Research Question 3 will be analyzed using survival analysis. We also used a Research-to-Practice Feedback Loop to catalyze rapid assessment of intervention and implementation refinement to increase participant responsivity.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Ages 18-35
* Have experienced at least one lifetime traumatic event
* Released from incarceration to Suwanee, Leon, Duval or Columbia County, Florida.
* Conversational in English
* Being able to cognitively consent

Exclusion Criteria:

* Younger than 18 years old
* Older than 35 years old
* Has not experienced at least one lifetime traumatic event
* Not cognitively able to understand
* Not conversational in English
* Not releasing from incarceration to Suwanee, Leon, Duval or Columbia County, Florida.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 403 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Pettus-Davis, PhD, Principal Investigator — Florida State University College of Social Work, Institute of Justice Research & Development; Stephen Tripodi, PhD, Principal Investigator — Florida State University College of Social Work, Institute of Justice Research & Development; Tanya Renn, PhD, Principal Investigator — Florida State University College of Social Work, Institute of Justice Research & Development
Locations (1):
- Institute for Justice Research and Development, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be considered for researchers and students, using the IJRD data sharing agreement. Data will be uploaded at the conclusion of the research to the National Archive of Criminal Justice Data, as required by the National Institute of Justice. Contact IJRD for additional information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be accessible for at least 6 years after the primary analyses have been published.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Started | 196 | 207
Completed | 28 (28 people completed 70% of programming) | 179 (179 people in the control group completed posttest and/or follow-up interviews.)
Not Completed | 168 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 196 | 207 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.07 (4.703) | 28.27 (4.664) | 28.17 (4.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 196 | 207 | 403
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 190 | 197 | 387
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 125 | 120 | 245
  White | 53 | 64 | 117
  More than one race | 13 | 19 | 32
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 196 | 207 | 403
BSI: Depression [Mean (Standard Deviation); unit: units on a scale] — Utilizing the Brief Symptom Inventory (BSI) to assess depression and anxiety symptoms in participants. The BSI is a 53-item self-report screening tool that asks respondents to rate their level of psychological distress over the past seven days based on a five-point Likert scale (0 = "not at all" to 5 = "extremely"). The BSI provides subscale scores on dimensions of somatization, depression, and anxiety as well as a Global Severity Index (GSI) that is calculated based on a sum of all items. Subscale scores range from 0 to 4. Higher scores on the BSI indicate higher levels of symptomology.
  units on a scale | .265 (.502) | .304 (.538) | .285 (.521)
BSI: Anxiety [Mean (Standard Deviation); unit: units on a scale] — Utilizing the Brief Symptom Inventory (BSI) to assess depression and anxiety symptoms in participants. The BSI is a 53-item self-report screening tool that asks respondents to rate their level of psychological distress over the past seven days based on a five-point Likert scale (0 = "not at all" to 5 = "extremely"). The BSI provides subscale scores on dimensions of somatization, depression, and anxiety as well as a Global Severity Index (GSI) that is calculated based on a sum of all items. Subscale scores range from 0 to 4. Higher scores on the BSI indicate higher levels of symptomology.
  units on a scale | .310 (.554) | .370 (.574) | .340 (.564)
Barratt Impulsivity Scale [Mean (Standard Deviation); unit: units on a scale] — Barratt Impulsivity Scale (BIS) assesses general impulsiveness on six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness). The BIS is composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Participants select a number on the following scale: 1 if you rarely or never act or think that way, 2 if you occasionally think that way, 3 if you often think that way, or 4 if you almost or always think that way. Scores range from 30 to 120. Population: Data missing on 24 participants due to data collection error.
  units on a scale
    number analyzed (Participants) | 181 | 196 | 377
    (all) | 63.45 (9.11) | 63.27 (9.79) | 63.36 (9.46)
BSI: Substance Use Disorder [Count of Participants; unit: Participants] — Utilizing the 9-item substance use disorder subscale of the MINI International Neuropsychiatric Interview (MINI) to assess current incidence of substance use disorders. Items are rated on a dichotomous Yes/No scale and follow psychiatric guidelines of the DSM-5.
  Participants
    Yes | 138 | 150 | 288
    No | 58 | 57 | 115
Coping Self-Efficacy: Problem-Focused Coping [Mean (Standard Deviation); unit: units on a scale] — CSES assess coping self-efficacy. 26-item self-report tool that asks respondents to indicate if they feel they can do accomplish 26 specific things if when they are having problems. Responses are based on an 10-point Likert scale. The CSES provides subscale scores on problem-focused coping, stopping unpleasant thoughts, and social support as well as a total coping score based on a sum of all items. Problem focused scores range from 0 to 60. Higher scores indicate higher levels of coping self-efficacy.
  units on a scale | 45.67 (8.25) | 44.14 (9.32) | 44.88 (8.84)
Coping Self-Efficacy: Stop Unpleasant Emotions and Thoughts [Mean (Standard Deviation); unit: units on a scale] — CSES assess coping self-efficacy. 26-item self-report tool that asks respondents to indicate if they feel they can do accomplish 26 specific things if when they are having problems. Responses are based on an 10-point Likert scale. The CSES provides subscale scores on problem-focused coping, stopping unpleasant thoughts, and social support as well as a total coping score based on a sum of all items. Stop Unpleasant Emotions and Thoughts scores range from 0 to 40. Higher scores indicate higher levels of coping self-efficacy.
  units on a scale | 30.28 (6.25) | 28.95 (7.06) | 29.59 (6.76)
Coping Self-Efficacy: Get Support from Family and Friends [Mean (Standard Deviation); unit: units on a scale] — CSES assess coping self-efficacy. 26-item self-report tool that asks respondents to indicate if they feel they can do accomplish 26 specific things if when they are having problems. Responses are based on an 10-point Likert scale. The CSES provides subscale scores on problem-focused coping, stopping unpleasant thoughts, and social support as well as a total coping score based on a sum of all items. Social support scores range from 0 to 30. Higher scores indicate higher levels of coping self-efficacy.
  units on a scale | 21.33 (5.77) | 20.75 (5.88) | 21.03 (5.82)
Ryff Psychological Well-Being: Autonomy [Mean (Standard Deviation); unit: units on a scale] — Ryff Psychological Wellbeing Index assesses participant wellbeing. Ryff is an 18-item self-report tool that asks respondents to indicate how strongly they agree with 18 statements. Responses are based on a seven-point Likert scale. Ryff provides subscale scores on dimensions of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance as well as a global wellbeing index that is calculated based on a sum of all items. Subscale scores range from 3 to 21 and the global wellbeing scores range from 18 to 126.
  units on a scale | 35.16 (3.76) | 35.07 (4.12) | 35.11 (3.94)
Ryff Psychological Well-Being: Environmental Mastery [Mean (Standard Deviation); unit: units on a scale] — Ryff Psychological Wellbeing Index assesses participant wellbeing. Ryff is an 18-item self-report tool that asks respondents to indicate how strongly they agree with 18 statements. Responses are based on a seven-point Likert scale. Ryff provides subscale scores on dimensions of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance as well as a global wellbeing index that is calculated based on a sum of all items. Subscale scores range from 3 to 21 and the global wellbeing scores range from 18 to 126.
  units on a scale | 32.38 (4.58) | 32.49 (4.91) | 32.44 (4.75)
Ryff Psychological Well-Being: Personal Growth [Mean (Standard Deviation); unit: units on a scale] — Ryff Psychological Wellbeing Index assesses participant wellbeing. Ryff is an 18-item self-report tool that asks respondents to indicate how strongly they agree with 18 statements. Responses are based on a seven-point Likert scale. Ryff provides subscale scores on dimensions of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance as well as a global wellbeing index that is calculated based on a sum of all items. Subscale scores range from 3 to 21 and the global wellbeing scores range from 18 to 126.
  units on a scale | 33.79 (3.88) | 33.97 (3.98) | 33.89 (3.93)
Ryff Psychological Well-Being: Relations to Others [Mean (Standard Deviation); unit: units on a scale] — Ryff Psychological Wellbeing Index assesses participant wellbeing. Ryff is an 18-item self-report tool that asks respondents to indicate how strongly they agree with 18 statements. Responses are based on a seven-point Likert scale. Ryff provides subscale scores on dimensions of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance as well as a global wellbeing index that is calculated based on a sum of all items. Subscale scores range from 3 to 21 and the global wellbeing scores range from 18 to 126.
  units on a scale | 32.43 (4.74) | 33.22 (4.38) | 32.84 (4.57)
Ryff Psychological Well-Being: Purpose in Life [Mean (Standard Deviation); unit: units on a scale] — Ryff Psychological Wellbeing Index assesses participant wellbeing. Ryff is an 18-item self-report tool that asks respondents to indicate how strongly they agree with 18 statements. Responses are based on a seven-point Likert scale. Ryff provides subscale scores on dimensions of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance as well as a global wellbeing index that is calculated based on a sum of all items. Subscale scores range from 3 to 21 and the global wellbeing scores range from 18 to 126.
  units on a scale | 34.53 (4.44) | 34.70 (3.63) | 34.62 (4.04)
Ryff Psychological Well-Being: Self-Acceptance [Mean (Standard Deviation); unit: units on a scale] — Ryff Psychological Wellbeing Index assesses participant wellbeing. Ryff is an 18-item self-report tool that asks respondents to indicate how strongly they agree with 18 statements. Responses are based on a seven-point Likert scale. Ryff provides subscale scores on dimensions of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance as well as a global wellbeing index that is calculated based on a sum of all items. Subscale scores range from 3 to 21 and the global wellbeing scores range from 18 to 126.
  units on a scale | 31.09 (5.00) | 30.68 (5.00) | 30.88 (5.00)

OUTCOME MEASURES:

1. Primary Outcome: Housing Stability
Description: Stable housing was defined as living in one's own room, apartment, or house, or with family, with an expected duration of residence of 4 months or more, or tenancy rights. A 10- item measure will assess housing stability.
Time Frame: 4 months post release
Population: Treatment group is treatment of the treated: Those who completed at least 70% of RISE programming.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Group: Completed at least 70 percent of RISE programming
- Control Group: Treatment As Usual
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 196 | 207
Participants
  Stable Housing | 17 | 65
  Not Housing Stable | 7 | 23
  Non-Responsive | 172 | 119

2. Primary Outcome: Housing Stability
Description: as for outcome 1
Time Frame: 8 months post release
Population: Treatment group is treatment of the treated: those who completed at least 70% of programming
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 196 | 207
Participants
  Stable | 18 | 60
  Not Housing Stable | 8 | 29
  Non-responsive | 170 | 118

3. Primary Outcome: Employment Stability
Description: Employment Stability is measure on a continuum, based on the number of jobs held in the last 4 months and number of days worked at each Employment. The employment must be for at least 15 hours a week. A 10-item measure will assess employment stability
Time Frame: 4 months post release
Population: Treatment group is treatment of the treated: Those who completed at least 70% of programming
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 196 | 207
Participants
  Employed | 16 | 67
  Not Employed | 7 | 18
  Non-Responsive | 173 | 122

4. Primary Outcome: Employment Stability
Description: Employment Stability is based on the number of jobs held in the last 4 months and number of days worked at each Employment. The employment must be for at least 15 hours a week. A 10-item measure will assess employment stability
Time Frame: 8 months post release
Population: Treatment group is treatment of the treated: Those who completed at least 70% or programming
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 196 | 207
Participants
  Employed | 22 | 69
  Not Employed | 4 | 18
  Non-Responsive | 170 | 120

5. Primary Outcome: Brief Symptom Inventory
Description: Utilizing the Brief Symptom Inventory (BSI) to assess depression and anxiety symptoms in participants. The BSI is a 53-item self-report screening tool that asks respondents to rate their level of psychological distress over the past seven days based on a five-point Likert scale (0 = "not at all" to 5 = "extremely"). The BSI provides subscale scores on dimensions of somatization, depression, and anxiety as well as a Global Severity Index (GSI) that is calculated based on a sum of all items. Subscale scores range from 0 to 4. Higher scores on the BSI indicate higher levels of symptomology.
Time Frame: 4 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 172 people excluded from the treatment group and 119 people excluded from the TAU control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 88
units on a scale | .451 (.804) | .536 (.813)

6. Primary Outcome: Brief Symptom Inventory
Description: as for outcome 5
Time Frame: 8 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 172 people excluded from the treatment group and 119 people excluded from the TAU control group. There were 172 people excluded from the treatment group and 119 people excluded from the TAU control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 88
units on a scale | .618 (.932) | .553 (.789)

7. Primary Outcome: Mini International Neuropsychiatric Interview
Description: Utilizing the 9-item substance use disorder subscale of the MINI International Neuropsychiatric Interview (MINI) to assess current incidence of substance use disorders. Items are rated on a dichotomous Yes/No scale and follow psychiatric guidelines of the DSM-5.
Time Frame: 4 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 167 people excluded from the treatment group and 118 people excluded from the TAU control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 29 | 89
Participants
  Substance Use Disorder | 8 | 22
  No Substance Use Disorder | 21 | 67

8. Secondary Outcome: Recidivism-violation
Description: Number of days to reincarceration for a technical violation.
Time Frame: 1 year post release
Reporting Status: Not Posted, anticipated posting 2025-11

9. Secondary Outcome: Recidivism-violation
Description: Number of days to reincarceration for a technical violation.
Time Frame: 2 year post release
Reporting Status: Not Posted, anticipated posting 2025-11

10. Secondary Outcome: Recidivism-violation
Description: Number of days to reincarceration for a technical violation.
Time Frame: 3 year post release
Reporting Status: Not Posted, anticipated posting 2025-11

11. Secondary Outcome: Recidivism-new Crime
Description: Number of days to reincarceration for a new crime.
Time Frame: 1 year post release
Reporting Status: Not Posted, anticipated posting 2025-11

12. Secondary Outcome: Recidivism-new Crime
Description: Number of days to reincarceration for a new crime.
Time Frame: 2 year post release
Reporting Status: Not Posted, anticipated posting 2025-11

13. Secondary Outcome: Recidivism-new Crime
Description: Number of days to reincarceration for a new crime.
Time Frame: 3 year post release
Reporting Status: Not Posted, anticipated posting 2025-11

14. Other Pre Specified Outcome: Depressive Symptoms
Description: Depressive symptoms marked by dysphoric mood, inactivity, lack of interest, insomnia, feelings of worthlessness, diminished ability to think, and thoughts of suicide. Depressive symptoms will be measured using the Brief Symptom Inventory, a 53-items with a 6 question sub-scale of depressive symptoms were a respondent characterizes the intensity of distress (0 ="not at all" to 4="extremely").The higher score the more depressive symptoms.
Time Frame: 8 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 170 people excluded from the treatment group and 117 people excluded from the TAU control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 90
score on a scale | .730 (.964) | .440 (.670)

15. Other Pre Specified Outcome: Anxiety Symptoms
Description: Anxiety symptoms identified as apprehension or fear of impending actual or imagined danger, vulnerability, or uncertainty. Anxiety Symptoms will be measured using the Brief Symptom Inventory is a 53-items with a 6 question sub-scale of anxiety symptoms were a respondent characterizes the intensity of distress (0 ="not at all" to 4="extremely").The higher score the more symptoms of anxiety.
Time Frame: 8 months post release
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 90
units on a scale | .60 (1.15) | .574 (.812)

16. Other Pre Specified Outcome: Incidence of Substance Use Disorder
Description: A pathological pattern of impairment related to the overuse of, or dependence on, psychoactive drugs, prescription medications, or other substances. A 9-item substance use disorder subscale of the MINI assesses current incidence of substance use disorders. Items are rated on a dichotomous Yes/No scale and follow psychiatric guidelines of the DSM-5.
Time Frame: 8 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 167 people excluded from the treatment group and 117 people excluded from the TAU control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 29 | 90
Participants
  Substance Use Disorder | 9 | 23
  No Substance Use Disorder | 20 | 67

17. Other Pre Specified Outcome: Coping Self-Efficacy Scale
Description: Utilizing the Coping Self-Efficacy Scale (CSES) to assess coping self-efficacy. The CSES is an 26-item self-report tool that asks respondents to indicate if they feel they can do accomplish 26 specific things if when they are having problems. Responses are based on an 11-point Likert scale (0 = "Cannot do at all" to 10 = "Certain can do"). The CSES provides subscale scores on dimensions of problem-focused coping, stopping unpleasant emotions and thoughts, and social support as well as a total coping self-efficacy score that is calculated based on a sum of all items. Problem focused subscale scores range from 0 to 60, emotion-focused subscale scores range from 0 to 40, and social support subscale scores range from 0 to 30. The total coping self-efficacy score ranges from 0 to 260. Higher scores indicate higher levels of coping self-efficacy.
Time Frame: 4 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 172 people excluded from the treatment group and 115 people excluded from the TAU control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 88
score on a scale
  Using Problem-Focused Coping | 45.58 (8.43) | 43.52 (13.45)
  Stop Unpleasant emotions and thoughts | 29.1667 (5.75339) | 29.4091 (9.03205)
  Get Support From Friends and Family | 20.1250 (5.47177) | 20.6818 (7.89812)

18. Other Pre Specified Outcome: Coping Self-efficacy
Description: he CSES is an 26-item self-report tool that asks respondents to indicate if they feel they can do accomplish 26 specific things if when they are having problems. Responses are based on an 11-point Likert scale (0 = "Cannot do at all" to 10 = "Certain can do"). The CSES provides subscale scores on dimensions of problem-focused coping, stopping unpleasant emotions and thoughts, and social support as well as a total coping self-efficacy score that is calculated based on a sum of all items. Problem focused subscale scores range from 0 to 60, emotion-focused subscale scores range from 0 to 40, and social support subscale scores range from 0 to 30. The total coping self-efficacy score ranges from 0 to 260. Higher scores indicate higher levels of coping self-efficacy.
Time Frame: 8 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 170 people excluded from the treatment group and 118 people excluded from the TAU control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 89
score on a scale
  Using Problem-Focused Coping | 48.23 (10.03) | 44.93 (10.16)
  Stop Unpleasant Emotions and Thoughts | 30.3462 (8.01470) | 29.0449 (8.76967)
  Get Support From Friends and Family | 18.3846 (7.46232) | 19.8764 (7.20767)

19. Other Pre Specified Outcome: Barratt Impulsivity Scale
Description: Utilizing the Barratt Impulsivity Scale (BIS) to assess general impulsiveness on six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and three second-order factors (attentional, motor, and non-planning impulsiveness). The BIS is composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Participants select a number on the following scale: 1 if you rarely or never act or think that way, 2 if you occasionally think that way, 3 if you often think that way, or 4 if you almost or always think that way. Scores range from 30 to 120. A higher score indicates greater impulsivity.
Time Frame: 4 months post release
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 88
score on a scale | 61.63 (8.49) | 61.63 (11.66)

20. Other Pre Specified Outcome: Barratt Impulsivity Scale
Description: as for outcome 19
Time Frame: 8 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 171 people excluded from the treatment group and 123 people excluded from the TAU control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Trauma-Based Reentry Program | Treatment as Usual (TAU)
Number analyzed (Participants) | 25 | 84
score on a scale | 59.96 (15.83) | 61.48 (12.93)

21. Other Pre Specified Outcome: Ryff Psychological Wellbeing Index
Description: Utilizing the Ryff Psychological Wellbeing Index to assess participant wellbeing. The Ryff is an 18-item self-report tool that asks respondents to indicate how strongly they agree or disagree with 18 statements. Responses are based on a seven-point Likert scale (1 = "strongly agree" to 7 = "strongly disagree"). The Ryff provides subscale scores on dimensions of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance as well as a global wellbeing index that is calculated based on a sum of all items. Subscale scores range from 3 to 21 and the global wellbeing scores range from 18 to 126. Higher scores indicate higher levels of wellbeing.
Time Frame: 4 months post release
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 24 | 88
score on a scale
  Autonomy: number analyzed (Participants) | 24 | 87
  Autonomy | 35.9538 (3.85023) | 33.0000 (4.77396)
  Environmental Mastery | 32.3333 (4.54606) | 31.0795 (5.69174)
  Personal Growth | 33.7917 (4.54905) | 33.2386 (4.39695)
  Positive Relations to Others: number analyzed (Participants) | 24 | 87
  Positive Relations to Others | 32.3043 (3.48288) | 31.6782 (6.16912)
  Purpose in Life | 35.2500 (3.57832) | 33.6705 (5.10065)
  Self-Acceptance: number analyzed (Participants) | 24 | 87
  Self-Acceptance | 32.5000 (3.40077) | 30.2529 (5.43721)

22. Other Pre Specified Outcome: Ryff Psychological Wellbeing Index
Description: as for outcome 21
Time Frame: 8 months post release
Population: Analysis of the comprehensive trauma-based reentry program is of those who completed at least 70% of programming and who participated in 4 month post release interviews. Analysis of the treatment group is of those who participated in post-release interviews. There were 170 people excluded from the treatment group and 119 people excluded from the TAU control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 26 | 88
score on a scale
  Autonomy: number analyzed (Participants) | 26 | 87
  Autonomy | 34.6538 (5.38102) | 34.2414 (5.11488)
  Environmental Mastery | 30.1154 (7.67503) | 31.1477 (6.34368)
  Personal Growth | 34.8077 (4.73303) | 34.0909 (5.52244)
  Positive Relations to Others | 31.2400 (6.51460) | 32.0568 (5.87486)
  Purpose in Life | 32.7692 (6.48264) | 33.5909 (5.24708)
  Self-Acceptance: number analyzed (Participants) | 26 | 86
  Self-Acceptance | 31.6800 (679902) | 30.5698 (6.69599)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: 0
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/207
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/207
Other Adverse Events (participants affected / at risk) | 0/196 | 0/207

LIMITATIONS AND CAVEATS:
The primary limitation is that there is a relatively small percentage of subjects in the treatment group that completed treatment, although this is a common limitation is reentry work.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04785677/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04785677/SAP_001.pdf
  • Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT04785677/ICF_002.pdf